CLINICAL TRIAL: NCT00409266
Title: CT Assessment of Minimally Invasive Surgery and Computer Assisted Navigation in Total Knee Arthropla
Brief Title: CT Assessment of Minimally Invasive Surgery and Computer Assisted Navigation in Total Knee Arthroplasty
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator medical practice didn't allow to move forward with the study.
Sponsor: Stryker Instruments (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NAV06-01US
Record Dates: First submitted 2006-12-06; First posted 2006-12-08 (Estimated); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Total Knee Arthroplasty

ARMS (1):
- Functional flexion axis of the knee (Other): The functional flexion axis of the knee can be established by computer-assisted intra-operative data, through range of motion techniques, not specific landmarks such as epicondyles.
  Interventions: Device: Computer assisted navigation

INTERVENTIONS:
Device: Computer assisted navigation

SUMMARY:
The functional flexion axis of the knee can be established by computer-assisted intra-operative data, through range of motion techniques, not specific landmarks such as epicondyles.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females over the age of 18 and equal to or less than the age of 60
* Patients scheduled for elective Total knee arthroplasty surgery
* Patients who have signed informed consent and HIPAA Authorization
* Able to speak and understand English

Exclusion Criteria:

* Patients presenting with evidence of recent trauma, active infection, chronic pain syndrome of the spine, dementia or have been diagnosed with Alzheimer's disease
* Pregnant women
* Patients that will not sign the informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2007-01 (Estimated); Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R S Oliver, M.D., Principal Investigator — Jordan Hospital
Locations (1):
- Jordan Hospital, Plymouth, Massachusetts, United States

REFERENCES:
- [Background] Stoeckl B, Nogler M, Krismer M, Beimel C, de la Barrera JL, Kessler O. Reliability of the transepicondylar axis as an anatomical landmark in total knee arthroplasty. J Arthroplasty. 2006 Sep;21(6):878-82. doi: 10.1016/j.arth.2005.10.020. PMID 16950043